CLINICAL TRIAL: NCT07040215
Title: The Effectiveness of Subacute Stroke Patients Receiving Robotic Assisted Gait Training
Brief Title: Effects on Subacute Stroke With Robotic Assistive Gait Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 250321
Record Dates: First submitted 2025-05-15; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Stroke Gait Rehabilitation
Keywords: physiotherapy; Robotic Assistive Gait Training
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional PT (Active Comparator): Conventional Physiotherapy
  Interventions: Other: Physiotherapy
- Robotic Gait Training (Experimental): Conventional Physiotherapy combined with Robotic Assistive Gait Training
  Interventions: Device: Freewalk lower limb Robotic Assistive Gait Training; Other: Physiotherapy

INTERVENTIONS:
Device: Freewalk lower limb Robotic Assistive Gait Training — Participants in this group will receive robotic-assisted gait training three times per week (every other day) for 30 minutes per session, using the FREE Walk exoskeleton device (FREE Bionics, Taiwan). The device assists with walking, standing, and sitting. A physical therapist will help the participant wear the exoskeleton and supervise the training, adjusting the level of robotic support and intensity based on the participant's ability. In addition to RAGT, participants will receive conventional stroke rehabilitation therapy (including sit to stand, balance and gait training) on the remaining weekdays (2 days/week), 30 minutes per session.
  Intervention Duration: 4 weeks.
  Arms: Robotic Gait Training
Other: Physiotherapy — Participants in this group will receive conventional stroke rehabilitation therapy (including sit to stand, balance and gait training) 5 days/week, 30 minutes per session. Intervention Duration: 4 weeks.

SUMMARY:
The goal of this randomized controlled trial is to learn about the effects of Robotic Assisted Gait Training (RAGT) combined with traditional physical therapy in subacute stroke patients. The main question it aims to answer is:

- Does RAGT combined with traditional physical therapy improve gait and functional performance in subacute stroke patients compared to traditional physical therapy alone? Participants who are subacute stroke patients will be randomly assigned to receive either both RAGT and traditional physical therapy or only traditional physical therapy. Their gait and functional performance will be assessed during the study period.

DETAILED DESCRIPTION:
The sequelae of stroke have a significant impact on patients' physical functions and quality of life. Although traditional physical therapy can help some patients regain function, its effectiveness is often limited. Therefore, exploring new rehabilitation technologies has become one of the key tasks in the medical field. Robotic Assisted Gait Training (RAGT) is an emerging technology that provides high-intensity and repetitive gait training, making it particularly suitable for patients in the post-stroke rehabilitation phase. Recent studies have shown that RAGT can significantly improve gait abilities in stroke patients, including walking speed and functional performance. Therefore, this study will adopt a randomized controlled trial design, recruiting 20 subacute stroke patients who will be randomly assigned to either a group receiving both RAGT and traditional physical therapy or a group receiving only traditional physical therapy. The study will compare differences in gait and functional performance between the two groups during the rehabilitation process, aiming to provide a foundation for future personalized and precision treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stroke (ischemic or hemorrhagic) confirmed by medical imaging.
* Subacute phase of stroke (onset within 1 to 3 months).
* Moderate to good standing balance ability.
* Sufficient cognitive ability to understand the study and follow instructions.
* Able to participate in rehabilitation training during the study period.

Exclusion Criteria:

* Body weight over 90 kg.
* Presence of other neurological disorders.
* Severe cardiovascular disease or other health conditions affecting mobility.
* Significant lower limb pain, joint contracture, or spasticity (Modified Ashworth Scale score > 3) that impairs walking.
* Diagnosed with cardiopulmonary disease that contraindicates exercise training.
* Cognitive impairment that prevents understanding of training instructions or completion of questionnaires.
* Inability to complete the rehabilitation training protocol.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Gait Speed | Baseline and after 4 weeks of intervention
  Gait speed will be calculated as distance divided duration. A timer will collect the duration (seconds, s) while subjects walk 3 meters (m, distance). The gait speed showed as (m/s) directly.
Step Length | Baseline and after 4 weeks of intervention
  Objective assessment of gait performance using two inertial sensors attached to the shoes. Measures include step length (meters)
Toe Clearance | Baseline and after 4 weeks of intervention
  Objective assessment of gait performance using two inertial sensors attached to the shoes. Measures include toe clearance (meters).
Timed Up and Go Test (TUG) | Baseline and after 4 weeks of intervention
  Assesses functional mobility and fall risk. Participants stand up from a chair, walk 3 meters, turn around, return, and sit down. The time taken to complete the task is recorded.
Functional Independence Measure (FIM) | Baseline and after 4 weeks of intervention
  Evaluates the level of a participant's independence in daily activities. The FIM includes 18 items across motor and cognitive domains, each scored from 1 (total assistance) to 7 (complete independence), with a total score range of 18 to 126.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | Baseline and after 4 weeks of intervention
  Assesses participants' static and dynamic balance abilities using a 14-item scale. Each item is scored from 0 to 4, with a total score ranging from 0 to 56. Higher scores indicate better balance.
30-Second Chair Stand Test (30-CST) | Baseline and after 4 weeks of intervention
  Measures lower limb strength and endurance. Participants are asked to stand up and sit down from a standard chair as many times as possible within 30 seconds, with arms crossed over the chest.
Surface Electromyography (sEMG) | Baseline and after 4 weeks of intervention
  Non-invasive recording of muscle activity during walking using adhesive electrodes placed on major lower limb muscles (e.g., quadriceps, tibialis anterior, gastrocnemius).
Short Form-12 Health Survey (SF-12) | Baseline and after 4 weeks of intervention
  Self-reported measure of health-related quality of life. Includes 12 questions covering 8 domains such as physical functioning, role limitations, pain, general health, vitality, social functioning, emotional role, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Su-Fen Liao, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No